CLINICAL TRIAL: NCT06472505
Title: Using Polyglycolic Acid Mesh Prevents Cerebrospinal Fluid Leakage: Clinical Application to Endoscopic Endonasal Transsphenoidal Surgery
Brief Title: Using Polyglycolic Acid Mesh Prevents Cerebrospinal Fluid Leakage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202011030DIPB
Record Dates: First submitted 2022-06-20; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Pituitary Tumor; Cerebrospinal Fluid Leakage
Keywords: Pituitary tumor; Endoscopic transnasal transsphenoidal; CSF leakage
MeSH Terms: conditions — Pituitary Neoplasms; Cerebrospinal Fluid Leak; Cerebrospinal Fluid Rhinorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Using polyglycolic acid mesh (Experimental)
  Interventions: Device: polyglycolic acid(Neoveil)

INTERVENTIONS:
Device: polyglycolic acid(Neoveil) — This study plans to enroll patients with pituitary tumors who need to undergo surgical treatment according to current routine medical standards. After the tumor tissue is removed, the integrity of the spider web or skull base will be thoroughly checked by endoscopy during the operation to confirm whether there is any cerebrospinal fluid leakage. At the end of the operation, use a 100*50*0.15mm, green sheet-like Navi tissue repair patch, cut it aseptically to fit the size of the defect for repair (the common case is 2*3.5cm defect), and place it on the spider web or skull base Tissue repair at the surgical site to prevent cerebrospinal fluid leakage.

SUMMARY:
The papers propose a new method to prevent postoperative cerebrospinal fluid leakage. Doctors use the absorbable polyglycolic acid (PGA) and fibrin glue to repair in surgery, prevent cerebrospinal fluid leakage and reduce the necessity of postoperative lumbar drainage after surgery. This study will analyze the changes in cerebrospinal fluid leakage in patients with pituitary tumors and skull base tumors after surgery, and further understand the effectiveness of Neoveil , as the basis for the development of new treatments.

DETAILED DESCRIPTION:
Neoveil, the main component, is polyglycolic acid (PGA), which is a kind of absorbable material, and is made into a soft and tension non-woven material by special processing with good tissue compatibility and degradability. In the human body, its strength will gradually decrease due to hydrolysis, and will eventually be absorbed and metabolized. In the process of absorption, at first its strength is reduced, then the mass will gradually decrease, and it will be completely absorbed after about 15 weeks. At present, the United States, Europe, Australia, China and South Korea have been marketed, it is applied to the spine , pituitary tumors , skull base tumors and aneurysm surgery,etc. inthe related field of Neurosurgery in foreign countries. It can prevent the leakage of cerebrospinal fluid, and reduce the postoperative hospital stay and the probability of complications after surgery. There is a license from the TFDA. In clinical, it can be used in the sutures of parts or fragile organs that do not need to be healed for a long time, such as the lung, liver, and digestive tract, by suture (thick slice and tube type) or adhesion (Sheet) In the tissue, it can strengthen the compressive ability of the local tissue, prevent the suture thread from splitting the suture tissue, prevent the lung tissue from leaking, reduce the blood and fluid leakage from the surgical site, and reduce the postoperative hospital stay and after the operation The complication rate .

ELIGIBILITY:
A. Inclusion criteria

1. Patients with primary or recurrent pituitary tumors require endoscopic nasal surgery.

B. Exclusion criteria

1. Patients with pituitary gland tumors who do not receive surgical treatment.
2. Patients with other brain tumors.
3. Patients allergic to polyglycolic acid (PGA).
4. Patients who have had previous radiation therapy or chemotherapy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mesurement CSF leakage grade change after surgery | 6 months
  Confirmation of change in CSF leakage grafe after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Abel Huang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan